CLINICAL TRIAL: NCT06316128
Title: EmploYEd Antithrombotic Therapies in Patients With Acute Coronary Syndromes HOspitalized in iTalian CCUs
Acronym: EYESHOT-2
Status: Completed | Type: Observational
Sponsor: Heart Care Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: K26
Record Dates: First submitted 2024-03-05; First posted 2024-03-18 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2024-06

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This registry has the aim to assess the use of different antithrombotic therapies, including untested drug combinations, routinely used during the hospitalization phase, with their timing, route and dose of administration, in consecutive patients discharged with a diagnosis NSTEMI or STEMI in Italian Cardiac care Units (CCUs) during a four-week study period.

DETAILED DESCRIPTION:
EYESHOT-2 is a prospective, multicenter, observational, nationwide survey of patients discharged with a diagnosis NSTEMI or STEMI admitted to Italian CCUs.

The survey will be designed to include all consecutive patients, who met the eligibility criteria, admitted in hospitals with or without cardiac catheterization laboratories and cardiac surgery facilities during a period of 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients aged 18 years or more, discharged with diagnosis of myocardial infarction (NSTEMI or STEMI) admitted to CCUs undergoing myocardial revascularization (PCI or CABG) or conservative treatment. At presentation, the diagnosis of NSTEMI will be based on the measurement of troponins and assessment of ECG changes, as suggested by European Society of Cardiology (ESC) guidelines; the diagnosis of STEMI will be characterized by an acute chest pain and persistent (>20 min) ST-segment elevation ≥ 1mm in two or more limb leads, or contiguous pre-cordial leads or left bundle branch block.
* Written informed consent signed. Patients who cannot provide the informed consent due to very severe clinical conditions can give their consent some hours/days after admission, when more favourable clinical conditions allow them to receive the appropriate information. Patients having died before giving informed consent may also be included unless the local Institutional Review Board (IRB) does not allow this procedure. In that case, it is strongly suggested to obtain relative(s) agreement through the collect of a signed informed consent.

Exclusion Criteria:

* Patients with a diagnosis of Unstable Angina,
* Patients developing MI after PCI or CABG,
* MI following non-cardiac surgery or traumatic causes,
* Patients with chest pain without elevation of troponin,
* Patients enrolled in Randomized Controlled Trial (RCTs),
* Patients already enrolled into the study from another CCU

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All consecutive patients, who met the eligibility criteria, admitted in hospitals with or without cardiac catheterization laboratories and cardiac surgery facilities during a period of 4 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 2806 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Antithrombotic therapies | 1 week
  The primary objective of the study is to describe at a national level the different antithrombotic therapies (alone or in combination) commonly employed from admission to discharge in NSTEMI or STEMI patients undergoing different therapeutic strategies (PCI, CABG, conservative). A particular focus will be given to antithrombotic therapies (combinations, timing of administration, indications) used (a) before PCI (pre-treatment) (b) in the cath lab during PCI [use of Glycoprotein IIb/IIIa inhibitors (GPIs), cangrelor, anticoagulants] and (c) during hospital stay.

OTHER OUTCOMES:
Assessment of in-hospital clinical events | 1 week
  An exploratory objective is the assessment of the rate of in-hospital clinical events (ischemic and hemorrhagic) in a large setting of NSTEMI or STEMI patients admitted to CCUs treated with different revascularization strategies and combinations of antithrombotic agents.

CONTACTS AND LOCATIONS:
Locations (189):
- Italy (189):
  - Ospedale Santo Spirito - Sc Cardiologia, Casale, AL
  - Ospedali Riuniti - Sod Cardiologia Ospedaliera E Utic, Ancona, AN
  - Irccs Inrca - Uo Cardiologia/Utic/Telecardiologia, Ancona, AN
  - Ospedale San Donato - U.O.C Cardiologia, Arezzo, AR
  - Ospedale Valdarno S. Maria Della Gruccia - U.O. Malattie Cardiovascolari, Montevarchi, AR
  - Aorn San Giuseppe Moscati - U.O. Cardiologia/Utic 'D. Rotiroti', Avellino, AV
  - Ospedale Miulli - U.O.C. Cardiologia - Utic, Acquaviva delle Fonti, BA
  - Ospedale Della Murgia - Fabio Perinei - S.C. Cardiologia-Utic, Altamura, BA
  - Ospedale San Paolo - Cardiologia-Utic, Bari, BA
  - Aou Policlinico - Uoc Cardiologia Ospedaliera, Bari, BA
  - Ospedale Di Venere - U.O.C. Di Cardiologia, Carbonara di Bari, BA
  - Ospedale Bolognini - Cardiologia E Unita' Coronarica, Seriate, BG
  - Ospedali Treviglio-Caravaggio - Cardiologia, Treviglio, BG
  - Ospedale Degli Infermi - Sc Di Cardiologia, Ponderano, BI
  - Presidio Ospedaliero "Santa Maria Del Prato" - U.O.C. Di Cardiologia-Utic, Feltre, BL
  - Ospedale Di Bentivoglio - U.O. Cardiologia Pianura, Bentivoglio, BO
  - Ospedale Maggiore - U.O.C. Di Cardiologia, Bologna, BO
  - Ospedale Policlinico S. Orsola-Malpighi - U.O. Cardiologia-Galie', Bologna, BO
  - Ospedale Perrino - U.O.C. Di Cardiologia, Brindisi, BR
  - Asst Spedali Civili - Cardiologia, Brescia, BS
  - Asst Franciacorta - Presidio Chiari - Cardiologia/Utic, Chiari, BS
  - Ospedale Di Desenzano Del Garda - Divisione Di Cardiologia - U.C.C., Desenzano del Garda, BS
  - Ospedale Civile 'La Memoria' - U.O. Di Cardiologia, Gavardo, BS
  - Istituto Clinico San Rocco - Unita' Operativa Di Cardiologia, Ome, BS
  - Ospedale Centrale Bolzano - Cardiologia E Prove Funzionali, Bolzano, BZ
  - Arnas G. Brotzu - Cardiologia Con Utic, Cagliari, CA
  - A.O.U. Cagliari Policlinico Monserrato - Sc Cardiologia Utic Emodinamica, Monserrato, CA
  - Ospedale A. Cardarelli - U.O. Cardiologia E Utic, Campobasso, CB
  - Presidio Ospedaliero Moscati - U.O.C. Cardiologia-Utic, Aversa, CE
  - Azienda Ospedaliera S. Anna E S. Sebastiano - U.O. Cardiologia D'Emergenza Con Utic, Caserta, CE
  - Casa Di Cura San Michele - Uo Cardiologia, Maddaloni, CE
  - Ospedale San Giuseppe E Melorio - U.O.C. Cardiologia Utic, Santa Maria Capua Vetere, CE
  - Presidio Ospedaliero San Rocco - U.O.C. Cardiologia - Utic, Sessa Aurunca, CE
  - Ospedale Policlinico Ss. Annunziata - Uoc Cardiologia-Utic, Chieti, CH
  - Azienda Ospedaliera Santa Croce E Carle - Sc Cardiologia, Cuneo, CN
  - Ospedale Pietro E Michele Ferrero - Cardiologia E Utic, Verduno, CN
  - Ospedale Moriggia Pelascini - Unita' Operativa Di Cardiologia, Gravedona, CO
  - Ospedale Maggiore - U.O. Cardiologia E Utic, Crema, CR
  - P.O. "Pugliese" - A.O.U. "Renato Dulbecco" - Utic-Emodinamica E Cardiologia Interventistica, Catanzaro, CZ
  - Ospedale M. Bufalini - U.O. Di Cardiologia-Utic, Cesena, FC
  - Ospedale G.B. Morgagni - L. Pierantoni - U.O. Cardiologia, Forlì, FC
  - Arcispedale Sant'Anna - U.O. Cardiologia, Ferrara, FE
  - Policlinico Riuniti - S.C. Di Cardiologia Universitaria-Utic, Foggia, FG
  - Ospedale Casa Sollievo Della Sofferenza - Cardiologia - Utic - Riabil Cardiologica, San Giovanni Rotondo, FG
  - Ospedale Santa Maria Annunziata - Sos Cardiologia Clinica, Bagno a Ripoli, FI
  - Ospedale San Giuseppe - Cardiologia, Empoli, FI
  - Ospedale Santa Maria Nuova - Cardiologia, Florence, FI
  - Aou Careggi - Interventistica Cardiologica Strutturale, Florence, FI
  - Ospedale Padre Antero Micone - Sc Cardiologia - Utic, Genova, GE
  - Ospedale Villa Scassi - Asl 3 Ligure - Sc Cardiologia Utic, Genova, GE
  - Ospedale Del Tigullio Polo Lavagna - Sc Cardiologia E Utic, Lavagna, GE
  - Presidio Ospedaliero - U.O. Cardiologia, Sanremo, IM
  - Ospedale Civile - S.C. Cardiologia, Ivrea, Ivrea
  - Ospedale San Leopoldo Mandic - Cardiologia - Ucc, Merate, LC
  - Ospedale Vito Fazzi - Uoc Cardiologia-Utic Ed Emodinamica, Lecce, LE
  - Ospedale Ignazio Veris Delli Ponti - Uoc Cardiologia-Utic "E. Vilei", Scorrano, LE
  - Azienda Osp. Cardinale G. Panico - U.O. Cardiologia - Utic, Tricase, LE
  - Ospedale Civile Bassa Val Di Cecina - Unita Operativa Di Cardiologia E Utic, Cecina, LI
  - Ospedali Riuniti - U.O.C. Cardiologia E Utic, Livorno, LI
  - Ospedale Villamarina - Cardiologia E Utic Piombino Elba, Piombino, LI
  - Ospedale Maggiore Di Lodi - U.O.C. Cardiologia, Lodi, LO
  - Nuovo Ospedale Versilia - Sc Cardiologia, Camaiore, LU
  - Ospedale Santa Croce - Uosd Cardiologia E Di Continuita Assist., Castelnuovo di Garfagnana, LU
  - Ospedale Pio Xi - U.O.C. Di Cardiologia, Desio, MB
  - Fondazione Irccs San Gerardo Dei Tintori - Ospedale San Gerardo - U.O.C. Cardiologia, Monza, MB
  - Nuovo Ospedale Di Vimercate - S.C. Cardiologia E Utic, Vimercate, MB
  - Presidio Osp. Di Civitanova Marche - Sc Cardiologia, Civitanova Marche, MC
  - Irccs Centro Neurolesi Bonino Pulejo - P.O. Piemonte - Cardiologia E Utic, Messina, ME
  - Humanitas Gavazzeni - U.O. Cardiologia, Bergamo, MI
  - Ospedale Di Cernusco Sul Naviglio - U. O. Di Cardiologia E Ucc, Cernusco sul Naviglio, MI
  - Ospedale Edoardo Bassini - Sc Cardiologia-Ucc Asst Nord Milano (Bassini-Ssg), Cinisello Balsamo, MI
  - Asst Ovest Milanese - Po Di Legnano - Cardiologia E Unita' Coronarica, Legnano, MI
  - Ospedale Civile Fornaroli - U.O. Cardiologia, Magenta, MI
  - Fondazione Irccs Ca' Granda Ospedale Maggiore Policlinico - Uoc Malattie Cardiovascolari, Milan, MI
  - Centro Cardiologico Monzino Irccs - Terapia Intensiva Cardiologica (Utic), Milan, MI
  - Ospedale San Luca Irccs - Istituto Auxologico - Area Critica Cardiologica, Milan, MI
  - ASST SANTI PAOLO E CARLO - PO San Carlo - CARDIOLOGIA-UCC, Milan, MI
  - Ospedale L. Sacco - Sc Cardiologia, Milan, MI
  - Asst Ospedale Metropolitano Niguarda - Cardiologia 1 - Emodinamica, Milan, MI
  - Ospedale Civile - Unita' Operativa Di Cardiologia, Rho, MI
  - Istituto Clinico Humanitas - Irccs - Cardiologia Clinica, Interventistica E Ucc, Rozzano, MI
  - Irccs Policlinico San Donato - U.O. Cardiologia Con Utic, San Donato Milanese, MI
  - Irccs Policlinico Multimedica - Uo Di Cardiologia, Sesto San Giovanni, MI
  - Ospedale Civile Di Baggiovara - U.O. Di Cardiologia, Modena, MO
  - Ospedale Di Sassuolo - Cardiologia, Sassuolo, MO
  - Ospedale Apuane - U.O. Cardiologia-Utic, Massa, MS
  - Ospedale Madonna Delle Grazie - Ssd Utic, Matera, MT
  - Ospedale San Francesco - Cardiologia - Utic, Nuoro, NU
  - Ospedale Giovanni Paolo Ii - Utic - Cardiologia, Olbia, OT
  - Fondazione G. Giglio - U.O. Di Cardiologia, Cefalù, PA
  - Aou Policlinico P. Giaccone - U.O.C. Cardiologia, Palermo, PA
  - Arnas P.O. Civico E Benfratelli - Uoc Utic, Palermo, PA
  - Ospedale G.F. Ingrassia - Cardiologia - Utic, Palermo, PA
  - Maria Eleonora Hospital - Cardiologia, Palermo, PA
  - Aor Villa Sofia-Cervello P.O. Cervello - U.O. Cardiologia - Cervello, Palermo, PA
  - Aor Villa Sofia-Cervello Po Villa Sofia - Uoc Cardiologia E Utic E Emodinamica -Villa Sofia, Palermo, PA
  - Ospedale Civile 'Guglielmo Da Saliceto' - Uoc Cardiologia E Utic, Piacenza, PC
  - Ospedale Civile Dello Spirito Santo - Cardiologia Con Utic, Pescara, PE
  - Presidio Ospedaliero Citta' Di Castello - U.O. Cardiologia/Utic, Città di Castello, PG
  - Nuovo Ospedale San Giovanni Battista - S.C. Cardiologia, Foligno, PG
  - Ospedale Gubbio-Gualdo Tadino - U.O. Di Utic E Cardiologia, Gubbio, PG
  - Azienda Ospedaliera Di Perugia - S.C. Cardiologia, Perugia, PG
  - Ftgm - Stabilimento Di Pisa - Cardiologia E Medicina Cardiovascolare, Pisa, PI
  - Ospedale Santo Stefano - U.O. Cardiologia, Prato, PO
  - Ospedale Civile - U.O.C. Cardiologia - Utic, Fidenza, PR
  - Azienda Ospedaliera Universitaria Parma - U.O.C. Di Cardiologia, Parma, PR
  - Ospedale Ss. Cosma E Damiano - Sos Cardiologia, Pescia, PT
  - Ospedale San Jacopo - Soc Cardiologia, Pistoia, PT
  - Presidio Ospedaliero San Salvatore - Cardiologia E Utic, Pesaro, PU
  - Fondazione Irccs Policlinico San Matteo - Uoc Cardiologia 1, Pavia, PV
  - Ospedale Civile - U.O. Di Cardiologia, Voghera, PV
  - Aor San Carlo - Ospedale San Carlo - Ssd Terapia Intensiva Cardiologica, Potenza, PZ
  - Ospedale Civile - Uo Servizio Cardiologia, Lugo, RA
  - Ospedale Civile Santa Maria Delle Croci - Uoc Cardiologia, Ravenna, RA
  - Grande Ospedale Metropolitano - Osp Riuniti Bianchi Melacrino - Uoc Cardiologia E Utic, Reggio Calabria, RC
  - Ospedale Civile Di Guastalla - Sos Cardiologia E Riabilitazione Card Area Nord, Guastalla, RE
  - Po Santa Maria Nuova - Ausl Re Irccs - Soc Cardiologia Ospedaliera, Reggio Emilia, RE
  - Ospedale Giovanni Paolo Ii - U.O.C. Cardiologia-Utic, Ragusa, RG
  - P.O. San Camillo de Lellis - U.O.C. Cardiologia, Rieti, RI
  - Ospedale Dei Castelli - U.O.C. Di Cardiologia E Utic, Ariccia, RM
  - European Hospital - U.O.C. Cardiologia Interventistica, Roma, RM
  - Ospedale San Camillo - Uoc Cardiologia, Roma, RM
  - Ospedale Sandro Pertini - Uoc Cardiologia, Roma, RM
  - Aurelia Hospital - U.O.C Cardiologia, Roma, RM
  - Policlinico Casilino - U.O.C. Cardiologia, Roma, RM
  - Ospedale Madre Giuseppina Vannini - U.O.C. Cardiologia, Roma, RM
  - Ospedale Isola Tiberina - Uoc Cardiologia Diagnostica Interventistica-Utic, Roma, RM
  - Ospedale Santo Spirito - Uoc Cardiologia, Roma, RM
  - Ospedale San Giovanni Evangelista - U.O.C. Di Cardiologia - Utic, Tivoli, RM
  - Ospedale Infermi - U.O. Cardiologia, Rimini, RN
  - Ospedale S. Maria Incoronata Dell'Olmo - U.O.C. Cardiologia-Utic, Cava de' Tirreni, SA
  - Ospedale Maria Ss. Addolorata - U.O. Di Cardiologia Utic, Eboli, SA
  - Presidio Ospedaliero Umberto I - Uoc Cardiologia - Utic, Nocera Inferiore, SA
  - Presidio Ospedaliero Luigi Curto - Uo Cardiologia-Utic, Polla, SA
  - Aou S. Giovanni Di Dio-Ruggi D'Aragona - Ssd Utic, Salerno, SA
  - Ospedale San Luca - U.O. Utic - Cardiologia, Vallo della Lucania, SA
  - Ospedale Dell'Alta Val D'Elsa - Uosd Cardiologia-Utic, Poggibonsi, SI
  - Aou Senese Ospedale S. Maria Alle Scotte - Cardiologia, Siena, SI
  - Ospedale S. Andrea - S.C. Cardiologia, La Spezia, SP
  - Ospedale E. Muscatello - U.O. Di Cardiologia - Utic, Augusta, SR
  - Ospedale G. Di Maria - Cardiologia Utic, Avola, SR
  - P.O. Lentini - Uosd Di Cardiologia Con Utic, Lentini, SR
  - Ospedale Ss. Annunziata - Cardiologia Clinica Ed Interventistica, Sassari, SS
  - Ospedale Nostra Signora Di Bonaria - U.O.C. Cardiologia E Utic, San Gavino Monreale, SU
  - Po Ponente - Ospedale Santa Corona - Sc Cardiologia Ponente, Pietra Ligure, SV
  - P.O. Levante - Ospedale San Paolo - S.C. Cardiologia Levante, Savona, SV
  - Ospedale Di Castellaneta - S.C. Cardiologia, Castellaneta, TA
  - Casa Di Cura Villa Verde - Cardiologia, Taranto, TA
  - Ospedale Ss. Annunziata - S.C. Cardiologia-Utic, Taranto, TA
  - Ospedale Santa Chiara - Divisione Di Cardiologia, Trento, TN
  - Ospedale Civico - Sc Cardiologia, Chivasso, TO
  - Por Cirie'- Lanzo Presidio Cirie' - S.C. Cardiologia, Cirié, TO
  - Ospedale Santa Croce - Cardiologia, Moncalieri, TO
  - Aou San Luigi Gonzaga - S.C.D.O. Cardiologia, Orbassano, TO
  - Ospedale Degli Infermi - Sc Cardiologia, Rivoli, TO
  - Aou Citta' Della Salute E Della Scienza - S.C. Cardiologia U, Torino, To
  - Ospedale Mauriziano Umberto I - Sc Cardiologia, Torino, TO
  - Ospedale Martini - Cardiologia (Mrt-Mv), Torino, TO
  - Ospedale Maria Vittoria - Cardiologia (Mrt-Mv), Torino, TO
  - Ospedale San Giovanni Bosco - Sc Cardiologia, Torino, TO
  - Po S. Antonio Abate Di Trapani - U.O.C. Di Cardiologia, Utic Ed Emodinamica, Erice, TP
  - Osp Abele Ajello - U.O.C. Cardiologia Con Utic, Mazara del Vallo, TP
  - Ospedale San Valentino - U.O.C. Cardiologia, Montebelluna, TV
  - Ospedale Ca' Foncello - U.O.C. Cardiologia, Treviso, TV
  - Pou "Santa Maria Della Misericordia" - S.O.C. Cardiologia, Udine, UD
  - Presidio Ospedaliero Di Saronno - U.O.C. Di Cardiologia, Saronno, VA
  - Ospedale San Biagio - Soc Cardiologia Vco, Domodossola, VB
  - Ospedale Castelli - Soc Cardiologia Vco, Verbania, VB
  - Ospedale Dell'Angelo - U.O.C. Cardiologia, Mestre, VE
  - Presidio Ospedaliero Di Mirano - U.O.C. Di Cardiologia, Mirano, VE
  - Ospedale Civile - U.O.C. Di Cardiologia, San Donà di Piave, VE
  - Ospedale Civile - U.O.C. Di Cardiologia, Arzignano, VI
  - Ospedale Civile San Bortolo - U.O.C. Cardiologia, Vicenza, VI
  - Ospedale G. Fracastoro - U.O.C. Di Cardiologia, San Bonifacio, VR
  - Aoui Di Verona - U.O. Cardiologia, Verona, VR
  - Ospedale Belcolle - Uosd Utic Polo, Viterbo, VT
  - Ospedale Ss. Trinita' - S.C. Di Cardiologia, Borgomanero
  - Ospedale Civile Di Boscotrecase - Utic Cardiologia, Boscotrecase
  - Ospedale San Leonardo - U.O. Di Cardiologia-Utic, Castellammare di Stabia
  - Ospedale San Giovanni Di Dio - Uo Cardiologia - Utic, Frattamaggiore
  - Presidio Ospedaliero San Giugliano - U.O. Cardiologia - Utic, Giugliano in Campania
  - Ospedale Anna Rizzoli - Cardiologia-Utic, Lacco Ameno
  - Aorn Cardarelli - U.O. Cardiologia Con Utic, Napoli
  - Aorn Ospedale Dei Colli - P.O. Monaldi - Uoc Cardiologia-Utic, Napoli
  - Ospedale Dei Pellegrini - Uoc Cardiologia-Utic, Napoli
  - Ospedale Del Mare - U.O. Cardiologia Con Utic-Emodinamica, Napoli
  - Pres. Ospedaliero S. Maria Della Pieta' - U.O. Cardiologia E Utic, Nola
  - Aou Maggiore Della Carita' - Scdo Cardiologia Ii, Novara
  - Ospedale Santa Maria Delle Grazie - U.O. Cardiologia - Utic Con Emodinamica, Pozzuoli

REFERENCES:
- [Result] Zuin M, Lucci D, Calabro P, Nicosia A, Tizzani E, Mauro C, Temporelli PL, Gonzini L, Maggioni AP, Grimaldi M, Colivicchi F, Gabrielli D, Oliva F, De Luca L. Acute pharmacologic management of myocardial infarction in patients undergoing percutaneous coronary intervention: insights from the Italian nationwide EYESHOT-2 prospective registry. Eur Heart J Open. 2025 Nov 25;5(6):oeaf154. doi: 10.1093/ehjopen/oeaf154. eCollection 2025 Nov. PMID 41377093
- [Result] De Luca L, Maggioni AP, Cavallini C, Leonardi S, Lucci D, Sacco A, di Uccio FS, Valente S, Navazio A, Pascale V, Geraci G, Lanni F, Gulizia MM, Colivicchi F, Gabrielli D, Oliva F; EYESHOT-2 Investigators. Clinical profile and management of patients with acute myocardial infarction admitted to cardiac care units: The EYESHOT-2 registry. Int J Cardiol. 2025 Jan 1;418:132601. doi: 10.1016/j.ijcard.2024.132601. Epub 2024 Sep 28. PMID 39349282